CLINICAL TRIAL: NCT06343597
Title: Volume Outcome Relationships and Effects of Adjuvant and Neoadjuvant Therapy in Mortality in Esophageal Cancer
Brief Title: Volume Outcome Relationships and Effects
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Methodist Health System (Other)
Responsible Party: Sponsor
Other Study IDs: 037.HPB.2020.R
Record Dates: First submitted 2022-04-27; First posted 2024-04-02 (Actual); Last update posted 2024-04-02 (Actual); Status verified 2023-04

CONDITIONS: Esophageal Cancer
MeSH Terms: conditions — Esophageal Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This is a retrospective analysis to assess if high-volume hospital facilities experience greater or lesser rates of incidence in patients with esophageal cancer than low-volume facilities.

DETAILED DESCRIPTION:
This is a retrospective analysis to assess if high-volume hospital facilities experience greater or lesser rates of incidence in patients with esophageal cancer than low-volume facilities.

The relationship between volume and outcomes has been proven in pancreatic cancer. Similar to pancreatic cancer, esophageal cancer historically has a bad prognosis. Esophageal cancer is typically asymptomatic, resulting in an advanced stage at the time of diagnosis. Additionally, it also has a significantly high morbidity and mortality. Therefore, it is crucial to determine volume-outcome relationships in esophageal cancer. This study aims to elucidate what these findings may entail by evaluating the impact that the volume-outcome relationship has on treatment assessment in esophageal cancer patients.

The purpose of the study is to evaluate the outcomes of esophageal cancer resection in patients in high volume (more than 5 esophagectomy performed per year) and low volume (less than 5 esophagectomy performed per year) hospital facilities. Furthermore, this paper will assess the outcomes of neoadjuvant and adjuvant therapy in esophageal cancer.

ELIGIBILITY:
Inclusion Criteria:

* esophageal cancer

Exclusion Criteria:

* No esophageal cancer

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: The purpose of the study is to evaluate the outcomes of esophageal cancer resection in patients in high volume (more than 5 esophagectomy performed per year) and low volume (less than 5 esophagectomy performed per year) hospital facilities.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2020-06-15 (Actual); Primary Completion 2025-06-15 (Estimated); Study Completion 2025-06-15 (Estimated)

PRIMARY OUTCOMES:
Esophageal Cancer resection in patients in high volume (more than 5 esophagectomy performed per year) and low volume (less than 5 esophagectomy performed per year) hospital facilities | through study completion, up to 18 months
  Retrospective analysis to assess if high-volume hospital facilities experience greater or lesser rates of incidence in patients with Esophageal Cancer than low-volume facilities

CONTACTS AND LOCATIONS:
Overall Officials: Dhiresh Jeyarajah, MD, Principal Investigator — Methodist Health System
Locations (1):
- Methodist Richardson Medical Center, Richardson, Texas, United States